CLINICAL TRIAL: NCT02372877
Title: Evaluation of the AMICUS Red Blood Cell Exchange (RBCx) System in Sickle Cell Patients
Brief Title: Evaluation of the AMICUS RBCx System in Sickle Cell Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenwal, Inc. (Industry)
Collaborators: Versiti Blood Health (Other); Children's Hospital of Philadelphia (Other); Barbara Ann Karmanos Cancer Institute (Other); University of Texas (Other); Washington University School of Medicine (Other); Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMIC-003-CMD
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle Cell Disease; Hemoglobin (Hb) S Disease; Hb S Disease; Congenital Hemolytic Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amicus Red Cell Exchange in SCD patients (Experimental): Open arm. Patients with sickle cell disease (SCD) treated using one Amicus Red Cell Exchange procedure.
  Interventions: Device: Amicus Red Cell Exchange in SCD patients

INTERVENTIONS:
Device: Amicus Red Cell Exchange in SCD patients — Each patient will be treated with one RBCx procedure using the AMICUS RBCx System
  Other Names: AMICUS RBCx System

SUMMARY:
The purpose of this study is to evaluate the performance of the AMICUS Red Blood Cell Exchange (RBCx) System (Exchange and Depletion/Exchange procedures) in patients with sickle cell disease.

DETAILED DESCRIPTION:
The goal of Red Blood Cell Exchange is to remove a patient's red blood cells (RBCs) and replace the blood volume removed with either healthy donor RBCs and/or colloid/crystalloid solutions. Depending on the RF used, the procedure can be considered an RBC Exchange or RBC Depletion/Exchange procedure. The RBC Depletion/Exchange procedure is a modification of the RBC Exchange procedure. The AMICUS RBCx protocol provides the ability to use various RFs including healthy donor RBCs or a combination of fluids, such as saline followed by RBCs. In RBC Exchange and the exchange portion of the RBC Depletion/Exchange procedures, RBC units are used as the RF, while colloid and/or crystalloid solutions are used as the RF in the depletion portion of the RBC Depletion/Exchange procedures. A new operating protocol on the AMICUS Separator that enables the device to perform Red Blood Cell Exchange (RBCx) procedures in accordance with the replacement fluid(s) (RF) prescribed by a physician for patients with sickle cell disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented diagnosis of a type of sickle cell disorder who require RBC Exchange or RBC Depletion/Exchange treatment.
* Medically stable subjects who have been previously treated for sickle cell disease with RBC Exchange or RBC Depletion/Exchange.
* Subjects, or subject's legal representative, who have provided signed informed consent, and assent when applicable, prior to participation.
* Adequate availability of sickle trait negative, leukoreduced, Blood type (ABO) blood group, Rhesus factor D (Rh (D)) compatible, unexpired replacement RBC products.
* Subjects with sufficient vascular access to accommodate the RBCx procedure as determined by the medical staff responsible for obtaining intravenous access.
* Subjects who are able and agree to report adverse events (AEs) during the required reporting period.

Exclusion Criteria:

* Procedures that occur during acute hospitalization.
* Procedures prescribed within one week of discharge of a hospitalization.
* Subjects with altered mental status that would prohibit the giving and understanding of informed consent, and assent when applicable, who do not have a legally authorized representative.
* Drug abuse, alcohol abuse, or other factors that in the opinion of the investigator could affect the ability of the subject to comply with the requirements of the protocol.
* Subjects who have experienced a serious adverse event associated with an RBCx procedure in the past.
* In the opinion of the investigator, subjects who have a life expectancy fewer than 30 days.
* Subjects who refuse blood products.
* Subjects who are pregnant.
* Subjects who fail to comply with site requirements for cessation of medication that interfere or increase procedure risk.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swerdlow, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (6):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amicus Red Cell Exchange or Depletion/Exchange in SCD Patients: Single-arm, open label study in patients with sickle cell disease (SCD) . SCD patients meeting the eligibility requirements will be treated with one RBCx procedure (Exchange or Depletion/Exchange) using the AMICUS RBCx System.
  The RBC Exchange or RBC Depletion/Exchange will be completed based on the physician's prescription.
Period: Overall Study
Arm/Group | Amicus Red Cell Exchange or Depletion/Exchange in SCD Patients
Started | 83
Completed | 59
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 63
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 80
  White | 0
  More than one race | 0
  Unknown or Not Reported | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83
Age at Procedure [Mean (Standard Deviation); unit: years] | 26.8 (10.26)

OUTCOME MEASURES:

1. Primary Outcome: Actual Fraction of Original Red Blood Cells Remaining to the Target Fraction of Cells Remaining (FCR).
Description: The primary endpoint will evaluate the mean ratio of the Actual FCR (FCRa) to Target FCR (FCRt) as measured by the patient's Hb S pre-procedure and post-procedure. The predefined mean ratio of the FCRa to FCRt is 0.75 to 1.25.
Time Frame: Actual FCR will be assessed by taking a pre-procedure sample from the patient on the day of the procedure and a post-procedure sample approximately 10-15 min after procedure completion.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 59
Ratio | 0.978 (.1933)

2. Secondary Outcome: Accuracy of Patient's End Hematocrit as Measured by the Patient's Post-procedure Hematocrit.
Description: Evaluate the accuracy of subject hematocrit post-procedure (End Hematocrit) (as measured by the patient's hematocrit at the end of the procedure) compared to the target End Hematocrit.
Time Frame: Actual End Hematocrit will be measured by taking a sample from the patient approximately 10-15 min after procedure completion.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 59
Ratio | 1.19 (0.817)

3. Secondary Outcome: Subject Cell Loss Post-Procedure (WBC)
Description: WBC loss post-procedure as measured with a complete blood count
Time Frame: Patient's blood cells will be measured by taking a sample from the patient approximately 10-15 min after procedure completion.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 59
Percentage of cells | 27.414 (21.6834)

4. Secondary Outcome: Serious Adverse Events
Description: Evaluate the number of device related serious adverse events during the procedure and approximately 18-24 hours post-procedure.
Time Frame: During the procedure up to 24 hours post-procedure.
Measure: Number; unit: Device Related Serious Adverse Events
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 83
Device Related Serious Adverse Events | 0

5. Secondary Outcome: Subject Cell Loss Post-Procedure (Platelets)
Description: Platelet loss post-procedure as measured with a complete blood count
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Amicus Red Cell Exchange in SCD Patients
Number analyzed (Participants) | 59
Percentage of cells | 48.967 (12.2895)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the procedure and 24 hours post-procedure.
Arm/Group | Amicus Red Cell Exchange in SCD Patients
All-Cause Mortality (participants affected / at risk) | 0/83
Serious Adverse Events (participants affected / at risk) | 2/83
Other Adverse Events (participants affected / at risk) | 12/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amicus Red Cell Exchange in SCD Patients (N=83)
Post Procedure - chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amicus Red Cell Exchange in SCD Patients (N=83)
During Procedure - Dizziness (Nervous system disorders) | 3 (3)
During Procedure - Device occlusion (General disorders) | 2 (2)
During Procedure - Chest Pain (General disorders) | 1 (1)
During Procedure - Vision blurred (Eye disorders) | 1 (1)
During Procedure - Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
During Procedure - Nausea (Gastrointestinal disorders) | 1 (1)
During Procedure - Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
During Procedure - Hypersensitivity (Immune system disorders) | 1 (1)
During Procedure - Blood pressure decreased (Investigations) | 1 (1)
During Procedure - Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
During Procedure - Catheterisation venous (Surgical and medical procedures) | 1 (1)
Post-Procedure - dizziness (Nervous system disorders) | 5 (5)
Post-Procedure - Headache (Nervous system disorders) | 1 (1)
Post-Procedure - Restless Legs Syndrome (Nervous system disorders) | 1 (1)
Post-Procedure - Nausea (Gastrointestinal disorders) | 2 (2)
Post-Procedure - Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Post-Procedure - Vomiting (Gastrointestinal disorders) | 1 (1)
Post-Procedure - Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Post-Procedure - back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Post-Procedure - fatigue (General disorders) | 1 (1)
Post-Procedure - Infusion site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post-Procedure - Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations or caveats apply to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02372877/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02372877/SAP_001.pdf